CLINICAL TRIAL: NCT03461458
Title: A Phase I Study Evaluating the Safety and Feasibility of Autologous, Culture-Expanded Adipose-Derived Mesenchymal Stromal Cells in Subjects With Painful Degenerative Disc Disease
Brief Title: Autologous, Culture-Expanded Mesenchymal Stromal Cells for Degenerative Disc Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator transition
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wenchun Qu, M.D., M.S., Ph.D., Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-002136
Record Dates: First submitted 2018-02-13; First posted 2018-03-12 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Degenerative Disc Disease
Keywords: Degenerative Disc Disease; Musculoskeletal Diseases; Lumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5×10^6 AD-MSCs (Experimental): Subjects will receive one injection of 5 million Autologous Adipose-Derived Mesenchymal Stromal Cells
  Interventions: Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells
- 20×10^6 AD-MSCs (Experimental): Subjects will receive one injection of 20 million Autologous Adipose-Derived Mesenchymal Stromal Cells
  Interventions: Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells

INTERVENTIONS:
Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells — Human, autologous, culture expanded, adipose-derived, mesenchymal stromal cells (AMSCs) produced on site in the Mayo Clinic Immune Progenitor and Cell Therapeutics Laboratory using current good manufacturing practices (cGMPs).
  Other Names: AMSCs

SUMMARY:
To determine the safety and feasibility of autologous, culture-expanded adipose-derived (AD) mesenchymal stromal cells (MSCs) in subjects with painful degenerative disc disease (DDD).

DETAILED DESCRIPTION:
This study is a prospective, phase I dose-escalation study evaluating the safety and feasibility of intradiscally injected AD-MSCs in the treatment of painful degenerative disc disease. The investigators propose a blended open enrollment protocol of four cohorts, each comprised of 3 subjects, to allow for interim analysis following the completion of each cohort to review safety data prior to commencing treatment of the next cohort. A total of 12 subjects will be enrolled. Subjects will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained baseline values will be established and subjects will begin treatment and follow-up for the next 24 months. Baseline data will include physical examination of the axial skeleton and sacroiliac region, neurologic examination, clinical assessment of low back pain and function using validated Patient Reported Outcome Measures (PROMs), radiographs, peripheral blood analysis, and MRI imaging.

Abdominal fat will be harvested through a small incision and processed by the Mayo Clinic IMPACT laboratory using current Good Manufacturing Practices (cGMPs) and previously established standard operating procedures (SOPs) to produce clinical grade, autologous, culture-expanded AD-MSCs for subsequent intradiscal injection. All injections will be performed using fluoroscopic guidance and all patients will be clinically evaluated immediately after procedure and at week 2 and 4 post-treatment to assess for acute adverse events (AEs). Following completion of their respective treatment cycle, each subject will be followed for study endpoints using a predetermined protocol, including clinical evaluation, radiography, MRI, and peripheral blood analysis. A final visit for evaluation and imaging will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age and older

   * Persons of childbearing potential must be non-nursing and have a negative serum pregnancy test prior to receiving the study drug and will agree to use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 24 months following completion of the drug treatment cycle. Persons of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using a kit.
   * Persons becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any serious adverse events (SAEs) associated with pregnancy will be recorded. The requirement for radiation (X-ray, MRI) will be removed.
2. Moderate radiographic degeneration of an Intervertebral Disc (IVD) from L1 to S1, with a disc suspected of causing chronic low back pain. Chronic low back pain is defined as the following:

   * Low back pain for at least 6 months
   * Failed at least 3 months of conservative back pain care. Conservative treatment regimens may include any or all of the following: initial rest, medications e.g., anti-inflammatory, analgesics, narcotics/opioids, muscle relaxants, massage, acupuncture, osteopathic or chiropractic manipulations, activity modification, home-directed lumbar exercise program, and non-invasive pain control treatments or procedures
   * Have at a minimum undergone supervised physical therapy, such as daily walking routines, therapeutic exercises, and back education programs specifically for the treatment of low back pain AND taken a pain medication for back pain (e.g. NSAID and/or opioid medication).
   * Low back pain of at least 30mm and not more than 90mm of 100mm on low back pain VAS (average pain over 24 hours)Radicular leg pain ≤20mm in both legs on a 100mm VAS scale
   * Oswestry Disability Index (ODI) score of at least 20 and no more than 90 on a 100 point scale.
3. Patients must demonstrate radiographic evidence of mild to moderate degenerative disc disease as defined by radiographic evidence of modified Pfirrmann scores of 3, 4, 5 or 6 on MRI at the index disc. With respect to inclusion criteria, DDD is defined as radiographic evidence of change from normal disc morphology of the index disc identified by modified Pfirrmann score and Modic Type I or II changes.

   • Change from normal disc morphology of the index disc will be determined based on radiographic evaluation. Radiographs must show all of the following as determined by participating fellowship trained radiologists at Mayo Clinic:
   * A modified Pfirrmann score of 3, 4, 5 or 6 on MRI at the index disc
   * Modic Grade II changes or less on MRI at the index disc
   * With or without contained disc protrusion at the index disc on MRI
4. Leg pain, if present, is of nonradicular origin, i.e., not due to stimulation of nerve roots or dorsal root ganglion of a spinal nerve by compressive forces.
5. Leg pain, if present, does not extend below the knee and is no greater than 50% of low back pain as measured on a visual analog scale. If bilateral leg pain is present, the worst leg pain is no greater than 50% of low back pain.
6. Full understanding of the requirements of the study and willingness to comply with the treatment plan, including laboratory tests, diagnostic imaging, and follow-up visits and assessments.
7. Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure.

Exclusion Criteria:

1. Subjects who are pregnant or nursing, or subjects planning to become pregnant in the first 24 months post-treatment. If a subject becomes pregnant during the study, the subject will remain in the study and only the requirement for radiation (x-ray or MRI) will be removed.
2. Extreme obesity, as defined by NIH Clinical Guidelines Body Mass Index (BMI > 40)
3. Have undergone a surgical procedure (e.g. discectomy, intradiscal electrothermal therapy, intradiscal radiofrequency, artificial disc replacement, interbody fusion) on the disc at the index or adjacent level
4. Osteoporosis, as defined by dual-energy X-ray absorptiometry (DEXA) scan. A DEXA T-score of ≤ -2.5 will exclude the subject. The following at-risk subjects will be required to undergo a DEXA scan at screening:

   1. Female subjects with a Simple Calculated Osteoporosis Risk Estimation (SCORE) of ≥6 and male subjects with a Male Osteoporosis Risk Estimation Score (MORES) of ≥6
   2. Females ≥50 years of age or who are post-menopausal or post-hysterectomy with oophorectomy
   3. Subjects taking bisphosphonate medications for the treatment of osteoporosis
   4. Subjects with a history of chronic, high-dose steroid use (oral and/or inhaled). High-dose steroid use is defined as:

   i. Daily, chronic use of oral steroids of ≥5 mg/day

   ii. Daily, chronic use of inhaled corticosteroids (at least twice per day)

   iii. Use of short-term (less than 10 days) oral steroids at a daily dose >20mg prednisone (or equivalent ) within 1 month of study procedure
5. Any lumbar intradiscal injection, including steroids, into the index or adjacent discs prior to treatment injection, with the exception of the following injections performed at least 2 weeks prior to study treatment:

   i. Contrast medium (discography or other diagnostic injection)

   ii. Nerve-blocking anesthetics (e.g., lidocaine, bupivacaine)

   iii. Antibiotics

   iv. Saline
6. Have undergone a procedure affecting the structure/biomechanics of the index disc level (e.g. posterolateral fusion)
7. Clinically relevant instability on flexion-extension as determined by the investigator by overlaying films.
8. Have an acute fracture of the spine at the time of enrollment in the study or clinically compromised vertebral bodies at the affected level due to current or past trauma, e.g., sustained pathological fracture or multiple fractures of vertebrae.
9. Presence of any of the following spinal deformities: scoliosis >10 degrees, spondylolysis at the index disc, spondylolisthesis > grade II at the index disc.
10. Presence of sequestered fragments, facet cysts, severe spinal stenosis, or severe disc degeneration at the index level and/or adjacent levels (as defined by modified Pfirrmann score greater than 6) by MRI.
11. Presence of a Grade V annular fissure on discography.
12. Presence of multi-level disc disease (> 1 level of involvement).
13. Epidural steroid injections within 8 weeks prior to treatment injection
14. Active malignancy or tumor as source of symptoms or history of malignancy within the 5 years prior to enrollment in study, except history of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or squamous cell carcinoma of the cervix if fully excised and with clear margins.
15. Currently participating in another investigational trial and/or plans to participate in any other allogeneic stem cell/progenitor cell therapy trial
16. Have been a recipient of prior allogeneic stem cell/progenitor cell therapy for any indication or autologous stem cell/progenitor cell therapy or other biological intervention to repair the index intervertebral disc
17. An average baseline morphine equivalent dose (MED) of >75mg/day, as determined by the investigator during Screening consultation.
18. Taking systemic immunosuppressant medications or having a chronic, immunosuppressive state.
19. Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment.
20. Clinically significant abnormal hematology (complete blood count with differential), blood chemistry, or urinalysis screening laboratory results, including aspartate aminotransferase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), bilirubin, creatinine, and C-Reactive Protein (CRP).
21. Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis.
22. Unexplained fever, defined as greater than 100.4 degrees Fahrenheit or 38.0 degrees Celsius, or mental confusion at baseline.
23. Clinically significant cardiovascular (e.g. history of myocardial infarction, congestive heart failure or uncontrolled hypertension > 90 mmHg diastolic and/or 180 mmHg systolic), neurologic (e.g. stroke, TIA) renal, hepatic, or endocrine disease (e.g. diabetes).
24. History of clinically significant blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy.
25. Participation in a study of an experimental drug or medical device within one year
26. Known allergy to local anesthetics of other components of the study drug.
27. Known history of hypersensitivity or anaphylactic reaction to murine or bovine products or dimethyl sulfoxide (DMSO).
28. Any contraindication to MRI according to MRI guidelines, or unwillingness to undergo MRI or X-ray procedures.
29. History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 30 days of study entry, as determined by the investigator during Screening consultation.
30. Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.
31. Being involved in active litigation related to subject's low back pain.
32. Have a mental illness that could prevent completion of the study or protocol questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience adverse events (AEs) | 2 years post final injection
  An adverse event is 1) Defined as any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline during the study regardless of causal relationship.

SECONDARY OUTCOMES:
Change in low back pain and function following injection of AD-MSCs | Baseline, treatment day, 2 weeks, 4 weeks, 3 months, 6 months, 12 months, 18 months, 24 months
  Change in low back pain will be measured by a 10 cm visual analog scale (VAS) score, with one end of the scale 0 indicating no pain, and the other end 10 indicating the worst pain ever.
Change in low back pain and function following injection of AD-MSCs | Baseline, treatment day, 2 weeks, 4 weeks, 3 months, 6 months, 12 months, 18 months, 24 months
  Change in low back pain and function will be measured by Global Health Scale (GHS) which includes health related questions with Likert Scales of 1 to 5, or 1 to 10. Based on the question, 1 may indicate a higher amount, or lower amount for the measured variable.
Change in low back pain and function following injection of AD-MSCs | Baseline, treatment day, 2 weeks, 4 weeks, 3 months, 6 months, 12 months, 18 months, 24 months
  Change in low back pain and function will be measured by Oswestry Disability Index (ODI), which contains 10 questions about daily activities with scores ranging from 0 to 5, where 0 indicates no difficulty/disability, and 5 indicates the most severe difficulty/disability. The final score is multiplied by 2 to give a final score from 0 to 100, where 0 is no difficulty/disability and 100 is severe difficulty/disability.
Change in low back pain and function following injection of AD-MSCs | Baseline, treatment day, 2 weeks, 4 weeks, 3 months, 6 months, 12 months, 18 months, 24 months
  Change in low back pain and function will be measured by Quality of Life (SF-36 questionnaire, which has questions regarding health and activity scored from 1 to 3, 1 to 5, or yes/no (1 to 2). Based on the question, 1 may indicate a lower amount/frequency or higher amount/frequency.
Change in low back pain and function following injection of AD-MSCs | Baseline, treatment day, 2 weeks, 4 weeks, 3 months, 6 months, 12 months, 18 months, 24 months
  Change in low back pain and function will be measured by Narcotic Use Questionnaire, which includes questions regarding the current use of narcotics (yes/no) and how long participants have used narcotics for pain relief (days, months, years).
Changes from Baseline in disc height index as measured by X-ray at 12 months and 24 months | Baseline, 12 Months, 24 Months
  An x-ray will be performed using standard radiography technology and interpreted by a trained radiologist.
Changes from Baseline in T2 weighted signal intensity of the Nucleus Pulposus (NP) as measured by MRI without contrast | Baseline, 6 Months, 12 Months, 24 Months
  Images will be obtained by MRI and interpreted by a trained radiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Wenchun Qu, MD, MS, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials